CLINICAL TRIAL: NCT01493609
Title: Computer Learning in Children - the Edinburgh Autism Social-attention Trial.
Brief Title: A Clinical Trial of a New Computer Based Intervention for Children With Autism.
Acronym: Click-East
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/C/PMLD/03; NCF/36343 (Other Grant/Funding Number: Nuffield Foundation)
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waitlist Control (No Intervention)
- Click-East app (Experimental): Participants will receive a copy of the game immediately following recruitment and assessment.
  Interventions: Behavioral: Click-East app

INTERVENTIONS:
Behavioral: Click-East app — Computer game, delivered as an iPad app, designed to provide an environment to practice basic social skills.
  Arms: Click-East app

SUMMARY:
The CLICK-EAST research project is an investigation of the efficacy of a computer based learning programme which aims to teach the fundamental components of social attention to young children with autism spectrum disorder (ASD). "Social attention" describes the process of choosing to look at or listen to social information in the world, normally in preference to any other available information. Social information normally refers to people: for example, we notice human voices more than birdsong or traffic noise, even if the latter is louder. As a rule, children with ASD are less likely to prioritise this kind of social information. This is thought to have a significant effect on their development and behaviour. For example, a child who doesn't listen to what his parents say may be very slow to learn language, and may also fail to follow important instructions. Our goal is to create a new learning programme, in the form of an enjoyable computer game, which encourages children to practise the skills of looking at and listening to people, despite the presence of distracting information. The investigators will develop the game with the input of an advisory group of parents and teachers of children with ASD as well as some young adults with an ASD diagnosis. Then they will perform a trial of the game with a group of preschoolers with ASD and their families, in order to determine whether the game is having a positive effect on the children's abilities.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of core autism
* aged between 15 months and 5 years, 11 months.
* minimum nonverbal age equivalent of 15 months.

Exclusion Criteria:

* Children with epilepsy whose developmental progress may be impeded
* families with little knowledge of the English language such that their understanding of the information sheets and instructions accompanying the trial is limited. Unfortunately funding is not available for the provision of translators or translated materials.

Ages: 15 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Autism Diagnostic Observation Schedule - Change (ADOS-C) | approx 6 months
  The primary outcome measure is the ADOS-C. The primary outcome will be: Is there a difference in ADOS-C composite score for children receiving the intervention compared to a treatment as usual control group? The ADOS-C is a detailed observation of social behaviours coded from the videoed interaction that takes place during the Autism Diagnostic Observation Schedule assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Fletcher-Watson, PhD, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - University of Edinburgh, Edinburgh, Midlothian
  - Clinical Research Facility, Royal Hospital for Sick Children, Edinburgh, Midlothian

REFERENCES:
- See also: Study website — http://www.dart.ed.ac.uk/click-east